CLINICAL TRIAL: NCT01186068
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Group Study of the Dose-Response Profile of V-101 Cream in Subjects With Erythematous Rosacea
Brief Title: Dose Response Study of Patients With Erythematous Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vicept Therapeutics, Inc. (Industry)
Collaborators: Accenture (Industry)
Responsible Party: Chief Operating Officer, Vicept Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V-101-ROSE-202
Record Dates: First submitted 2010-08-17; First posted 2010-08-20 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-08

CONDITIONS: Erythematous (Type One) Rosacea
Keywords: Rosacea, erythema
MeSH Terms: conditions — Rosacea; Erythema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- V-101 Cream 0.01% Concentration (Experimental): Low dose
  Interventions: Drug: V-101
- V-101 Cream 0.06% Concentration (Experimental): Mid-dose
  Interventions: Drug: V-101
- V-101 Cream 0.1% Concentration (Experimental): Mid-dose
  Interventions: Drug: V-101
- V-101 Cream 0.15% Concentration (Experimental): High dose
  Interventions: Drug: V-101
- Vehicle (Placebo Comparator): Cream without an active ingredient
  Interventions: Other: vehicle

INTERVENTIONS:
Drug: V-101 — Cream QD
  Arms: V-101 Cream 0.01% Concentration; V-101 Cream 0.06% Concentration; V-101 Cream 0.1% Concentration; V-101 Cream 0.15% Concentration
Other: vehicle — Cream QD
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the dose-response relationship (effect) of four concentrations of V-101 Cream in patients with erythematous(redness) rosacea.

DETAILED DESCRIPTION:
Patients must have moderate to severe erythematous (facial redness) rosacea

* Male and female patients must be at least 18 years old and in good general health
* Female patients must not be pregnant or nursing

ELIGIBILITY:
Inclusion Criteria:

* male or females at least 18 years of age
* diagnosis of stable erythematous rosacea
* < 3 inflammatory lesions
* in good general health
* females must be non-pregnant and non-lactating
* must be willing to sign a consent form

Exclusion Criteria:

* have ocular, phymatous or other types of rosacea
* allergy to any ingredient in study drug
* participation in other investigational studies within 30 days of enrollment
* use of systemic steroids within 28 days of Baseline
* use of tetracycline antibiotics within 28 days of baseline
* use of products containing oxymetazoline within 14 days of baseline
* use of topical steroids witin treatment area 14 days prior to baseline
* use of Rx or OTC products for treatment of acne or rosacea within 14 days of baseline
* use of any product for reducing redness within the treatment area witin 14 days prior to baseline
* use of monoamine oxidase (MAO) inhibitors
* use of niacin >/= 500mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2010-08

PRIMARY OUTCOMES:
Clinician's Erythema Assessment | Day 28 visit
  Physician visual evaluation

SECONDARY OUTCOMES:
Subject's Self Assessment | 28 Day Visit
  Patient assesses their condition

CONTACTS AND LOCATIONS:
Overall Officials: Stacy R Smith, MD, Principal Investigator — Therapeutics Clinical Research; Michael T Jarratt, MD, Principal Investigator — Derm Research, PLLC; Leslie S Baumann, MD, Principal Investigator — Baumann Cosmetic & Research Institute; Joseph F Fowler, MD, Principal Investigator — Dermatology Specialists Research; Robert T Matheson, MD, Principal Investigator — Oregon Medical Research Center, PC; Daniel M Stewart, DO, Principal Investigator — DBA Michigan Center for Skin Care Research; Eduardo Tschen, MD, Principal Investigator — Academic Dermatology Associates
Locations (7):
- United States (7):
  - Therapeutics Clinical Research, San Diego, California
  - Baumann Cosmetic & Research Institute, Miami Beach, Florida
  - Dermatology Specialists Research, Louisville, Kentucky
  - DBA Michigan Center for Skin Care Research, Clinton Twp, Michigan
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Oregon Medical Research Center, PC, Portland, Oregon
  - DermResearch, Inc., Austin, Texas